CLINICAL TRIAL: NCT01643122
Title: Validation Study to Assess Psychometric Properties of a Newly Developed Patient Reported Outcome Tool for Endometriosis
Brief Title: Validation Study for Endometriosis PRO
Acronym: VALEPRO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15849
Record Dates: First submitted 2012-07-04; First posted 2012-07-17 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Endometriosis
Keywords: Endometriosis, Validation study
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Other: No drug
- Group 2
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — Patients with expected stable endometriosis management status (EMS), i.e. patients who have not planned a change in endometriosis treatment or a therapeutic surgical procedure in the next 12 weeks and have had no change in endometriosis treatment or therapeutic surgical procedure in the previous 4 weeks.lease specify as free-text; for drugs include daily dose, dosage form dosage frequency and duration (if appl. and possible for the OS/NIS).
  Groups: Group 1
Other: No drug — Patients with expected change in endometriosis management status (EMS), i.e. patients who have planned a change in endometriosis treatment or a therapeutic surgical procedure during the next 12 weeks or have undergone a change in endometriosis treatment or a therapeutic surgical procedure in the previous 4 weeks.
  Groups: Group 2

SUMMARY:
Assess the psychometric properties of the Endometriosis Symptom Diary (ESD) and the Endometriosis Impact Scale (EIS) and provide evidence whether the PRO measures are reliable, valid and able to detect changes over time in approximately 250 patients with mild, moderate or severe endometriosis confirmed by laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Women with endometriosis confirmed by laparoscopy or laparotomy within five years before the baseline visit
* Good general health (except for findings related to endometriosis) as proven by medical history
* Patient has experienced endometriosis symptoms (i.e. pain) in the past 4 weeks, as assessed by a numerical rating scale (NRS)

Exclusion Criteria:

* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Undiagnosed abnormal genital bleeding
* Abuse of alcohol, drugs, or medicine (e.g., laxatives)
* Simultaneous participation in another clinical trial. Participation in another clinical trial prior to study entry that might have an impact on the study objectives, at the discretion of the investigator.
* Major surgery scheduled for the study period, except therapeutic surgical procedure for endometriosis
* Close affiliation with the study site; e.g. a close relative of the investigator, dependent person (e.g. employee or student of study site)
* Inability to cooperate with the study procedures for any reason, including the following examples: language comprehension, psychiatric illness, inability to get to the study site
* Previous enrollment to this study
* Regular use of pain medication due to other underlying diseases
* Known pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with endometriosis confirmed by laparoscopy
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Endometriosis symptoms rated by the Endometriosis Symptom Diary | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- United States (19):
  - Jonesboro, Arkansas
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - New Haven, Connecticut
  - Decatur, Georgia
  - Champaign, Illinois
  - Worcester, Massachusetts
  - Rochester, Minnesota
  - Brooklyn, New York
  - Greensboro, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - San Angelo, Texas
  - Salt Lake City, Utah
  - Sandy City, Utah
  - Norfolk, Virginia
  - Seattle, Washington
- Many Locations, Germany

REFERENCES:
- [Derived] Seitz C, Lanius V, Lippert S, Gerlinger C, Haberland C, Oehmke F, Tinneberg HR. Patterns of missing data in the use of the endometriosis symptom diary. BMC Womens Health. 2018 Jun 8;18(1):88. doi: 10.1186/s12905-018-0578-0. PMID 29884234